CLINICAL TRIAL: NCT04228562
Title: Consumer Motivation for Disease Prevention 2 (Clear Labels)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Yeung Wing Man, Associate Professor of Marketing, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 14507018(2)
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Factorial Assignment The study has a 2 (Factor: one modifiable cause vs. one modifiable + one non-modifiable causes) ✕ 2 (Anticipated regret induction: yes vs. no) between-subject design. Participants will be randomly assigned to one of the 4 between-subject conditions.
  There is also a within-subject variable. Each subject will respond to 10 rounds of decision task with 5 different levels of overall disease risk reduction brought by the removal of X. The 5 levels of risk reduction are: (i) Removal of X reduces disease risk from 60% to 50% ; (ii) 60% to 40%; (iii) 60% to 30%; (iv) 60% to 20%; (v) 60% to 10%.
Who Masked: Participant, Investigator
Masking Description: Each participant will only receive the instruction pertaining to the arm to which he/she is assigned. The Research Assistant who conducts the study does not know about the hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-modifiable factor ABSENT; NO anticipated regret induced (No Intervention): The experiment comprises 10 rounds of decision tasks. Participant begins with 130 points (each worth HK$0.5) in each round. After the 10 rounds, the computer randomly selects 1 round and the points from this round is paid in cash.
  There is a chance for the participant to develop a disease. Without prevention, the chance of getting the disease is 60%. A cause, X, is identified for the disease. X is a modifiable cause, which means that it can be changed by taking some actions. The participant has to decide whether or not to remove X. Removal of X reduces disease chance; the reduced chance varies between 10% and 50% across the 10 rounds and the exact level is communicated at the beginning of each round. The removal of X costs 30 points. Whether s/he ends up developing the disease or not is determined by a computerized lottery based on these chances. If s/he develops the disease, s/he will lose 100 points.
- Non-modifiable factor ABSENT; anticipated regret induced (Experimental): Same description as in the "uncontrollable factor absent, no anticipated regret induced" arm, except that the participants are induced to think to what extent they will feel regretful: a) if s/he decides not to remove X but ends up developing the disease and b) if s/he decides to remove X but still gets the disease.
  Interventions: Other: induction of anticipated regret
- Non-modifiable factor PRESENT; NO anticipated regret induced (Experimental): The experiment comprises 10 rounds of decision tasks. Participant begins with 130 points (each worth HK$0.5) in each round. After the 10 rounds, the computer randomly selects 1 round and the points from this round is paid in cash.
  There is a chance for the participant to develop a disease. Without prevention, the chance of getting the disease is 60%. Two causes, X and Y, are identified for the disease. X is a modifiable cause, which means that it can be changed by taking some actions. The participant has to decide whether or not to remove X. Removal of X reduces disease chance; the reduced chance varies between 10% and 50% across the 10 rounds and the exact level is communicated at the beginning of each round. The removal of X costs 30 points. Whether s/he ends up developing the disease or not is determined by a computerized lottery based on these chances. If s/he develops the disease, s/he will lose 100 points.
  Interventions: Other: non-modifiable factor
- Non-modifiable factor PRESENT; anticipated regret induced (Experimental): Same as the "uncontrollable factor present, no anticipated regret induced" arm, except that the participants are induced to think to what extent they will feel regretful: a) if s/he decides not to remove X but ends up developing the disease and b) if s/he decides to remove X but still gets the disease.
  Interventions: Other: non-modifiable factor; Other: induction of anticipated regret

INTERVENTIONS:
Other: non-modifiable factor — the presence of an uncontrollable / unremovable risk factor for a disease
  Arms: Non-modifiable factor PRESENT; NO anticipated regret induced; Non-modifiable factor PRESENT; anticipated regret induced
Other: induction of anticipated regret — higher level of elaboration on potential regret
  Arms: Non-modifiable factor ABSENT; anticipated regret induced; Non-modifiable factor PRESENT; anticipated regret induced

SUMMARY:
The purpose of this study is to examine (1) how the causal structure of a disease influences people's disease prevention decisions; and (2) how the causal structure of a disease interacts with people's regret anticipation in determining their disease prevention decisions.

DETAILED DESCRIPTION:
People sometimes have to deliberate on whether or not to remove a risk factor that may potentially cause a disease in the future. When a modifiable risk factor (say, X) is the only factor that causes a disease, the decision to remove it may simply depend on the probabilistic relationship between X and an outcome, as well as the cost of removing X. However, little is known when other factors that are out of the decision-maker's control are also present. The main question being asked here is how does the presence of such non-modifiable factors change people's decision to remove X.

Specifically, the investigators consider two cases: a disease caused by a single modifiable risk factor (say X) and a disease caused by two risk factors -- a modifiable factor (X) and a non-modifiable factor (Y). In both cases, the removal of X can result in a meaningful reduction in overall disease risk. It is hypothesized that even when the magnitude of overall risk reduction brought by the removal of X is the same in the two cases, people would have a lower motivation to remove X in the latter case.

The investigators also examine how the presence of a non-modifiable risk factor interacts with the respondents' regret anticipation to influence their decision to remove X. In the context of the current research, regret anticipation could take one of the following forms: (a) feel regretful if one decides not to remove X and later develops the disease (b) feel regretful if one decides to remove X but still develops the disease. The investigators expect (a) to moderate the effect of non-modifiable risk factor on motivation to remove X.

ELIGIBILITY:
Inclusion Criteria:

* students currently studying at the Chinese University of Hong Kong

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Decision to remove X | Day 1: When responding to the questionnaire
  The decision to remove X (yes vs. no)

OTHER OUTCOMES:
Anticipated regret | Day 1: When responding to the questionnaire
  The exact question is: Some people may engage in the following thoughts when they make their decisions: "I may regret if I do not remove X and end up getting the disease" OR "I may regret if I remove X but still get the disease." To what extent have you engaged in any of these thoughts? (Measurement scale: 1 = not at all; 7 = a lot)
Judgment of whether the removal of X is an opportunity to improve earnings | Day 1: When responding to the questionnaire
  The exact question is: Do you think the decision to remove X is an opportunity for you to improve your final earnings? (Measurement scale: 1 = not a good opportunity at all; 7 = a very good opportunity")
Sense of control over the final outcome | Day 1: When responding to the questionnaire
  The exact question is: Do you think you have control over the outcome through your decision of whether or not to remove X? (Measurement scale: 1 = I have very little control… 7 = I have a lot of control)

CONTACTS AND LOCATIONS:
Overall Officials: Wing Man Yeung, PhD, Principal Investigator — Chinese University of Hong Kong, Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to file sharing sites for sharing. Any identifying information will be removed before data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after manuscript is published, for 5 years starting from publication date.
Access Criteria: Data will only be made available for research purpose.

REFERENCES:
- [Background] Binder S, Nuscheler R. Risk-taking in vaccination, surgery, and gambling environments: Evidence from a framed laboratory experiment. Health Econ. 2017 Dec;26 Suppl 3:76-96. doi: 10.1002/hec.3620. PMID 29285871